CLINICAL TRIAL: NCT01589822
Title: A Single Blind, Randomized, Controlled Study to Evaluate the Safety and Effectiveness of EVICEL® as an Adjunct to Gastrointestinal Anastomosis Techniques
Brief Title: The EVICEL® Gastrointestinal Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 400-11-002
Record Dates: First submitted 2012-04-30; First posted 2012-05-02 (Estimated); Results first posted 2015-02-25 (Estimated); Last update posted 2015-02-25 (Estimated); Status verified 2015-02

CONDITIONS: Gastrointestinal Diseases
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- EVICEL Fibrin Sealant: Randomized (Experimental): EVICEL is a human plasma-derived fibrin sealant composed of two components - thrombin and fibrinogen.
  Interventions: Biological: EVICEL Fibrin Sealant
- Standard of Care (No Intervention): Standard surgical technique for GI anastomosis.
- Experimental: EVICEL Fibrin Sealant: Non-Randomized (Experimental): EVICEL is a human plasma-derived fibrin sealant composed of two components - thrombin and fibrinogen
  Interventions: Biological: EVICEL Fibrin Sealant

INTERVENTIONS:
Biological: EVICEL Fibrin Sealant — Intraoperative
  Other Names: Fibrin sealant
  Arms: EVICEL Fibrin Sealant: Randomized; Experimental: EVICEL Fibrin Sealant: Non-Randomized

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of EVICEL® Fibrin Sealant (Human) for use as an adjunct to gastrointestinal (GI) surgery.

DETAILED DESCRIPTION:
This is a single blind, randomized, multi-center controlled study evaluating the safety and effectiveness of EVICEL® when used as an adjunct to gastrointestinal (GI) surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing primary elective GI surgery
* Subjects ≥ 18 years of age who are willing to participate in the study and provide written informed consent prior to any study-related procedures

Exclusion Criteria:

* Avastin use within 30 days prior to surgery;
* Known hypersensitivity to the human blood products or the components of the investigational product;
* Female subjects who are pregnant or nursing;
* Exposure to another investigational drug or device in a clinical trial within 30 days prior to surgery or planned/intended for the 90 day follow up period after surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2012-06; Primary Completion 2014-01 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kocharian, MD, Study Director — Ethicon, Inc.
Locations (22):
- United States (8):
  - Clinical Investigation Site #1, Irvine, California
  - Clinical Investigation Site #2, Jacksonville, Florida
  - Clinical Investigation Site #5, Augusta, Georgia
  - Clinical Investigation Site #4, New Orleans, Louisiana
  - Clinical Investigation Site #8, Portland, Oregon
  - Clinical Investigation Site #23, Greenville, South Carolina
  - Clinical Investigation Site #3, Houston, Texas
  - Clinical Investigation Site #6, Houston, Texas
- Australia (2):
  - Clinical Investigation Site #19, New Lambton, New South Wales
  - Clinical Investigation Site #18, South Adelaide
- Belgium (2):
  - Clinical Investigation Site #17, Genk
  - Clinical Investigation Site #16, Ghent
- Canada (2):
  - Clinical Investigation Site #10, Vancouver, British Columbia
  - Clinical Investigation Site #9, Toronto, Ontario
- Clinical Investigation Site #20, Auckland, New Zealand
- South Korea (2):
  - Clinical Investigation Site #22, Seoul
  - Clinical Investigation Site #21, Seoul
- United Kingdom (5):
  - Clinical Investigation Site #15, Edinburgh
  - Clinical Investigation Site #11, Leicester
  - Clinical Investigation Site #12, Nottingham
  - Clinical Investigation Site #13, Plymouth
  - Clinical Investigation Site #14, Sheffield

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EVICEL Fibrin Sealant: Randomized | Standard of Care | Experimental: EVICEL Fibrin Sealant: Non-Randomized
Started | 84 | 89 | 41
Completed | 80 | 86 | 40
Not Completed | 4 | 3 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Missed 90 day visit | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Subjects enrolled who consented and were randomized into the study or assigned to the non-randomized portion and had the investigational product applied were included in the analysis sets. The Safety Set consists of 125 subjects treated with EVICEL (41 Non- Randomized) and 89 subjects treated with Standard of Care.
Groups:
- Total: Total of all reporting groups
Arm/Group | EVICEL Fibrin Sealant: Randomized | Standard of Care | Experimental: EVICEL Fibrin Sealant: Non-Randomized | Total
Number analyzed (Participants) | 84 | 89 | 41 | 214
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (11.1) | 62.5 (10.8) | 62.0 (12.2) | 61.8 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 33 | 21 | 95
  Male | 43 | 56 | 20 | 119
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 21 | 21 | 8 | 50
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 61 | 65 | 31 | 157
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 15 | 17 | 13 | 45
  Canada | 2 | 2 | 4 | 8
  Belgium | 17 | 17 | 3 | 37
  Australia | 10 | 9 | 6 | 25
  New Zealand | 10 | 10 | 1 | 21
  United Kingdom | 10 | 14 | 7 | 31
  Korea, Republic of | 20 | 20 | 7 | 47

OUTCOME MEASURES:

1. Primary Outcome: Absence of Gastrointestinal (GI) Leak
Time Frame: 40 days
Measure: Number; unit: participants
Groups:
- EVICEL Fibrin Sealant: Randomized: EVICEL is a human plasma-derived fibrin sealant composed of two components - thrombin and fibrinogen.
  EVICEL Fibrin Sealant: Intraoperative (IIT)
- Standard of Care: Standard surgical technique for GI anastomosis. (IIT)
- Experimental: EVICEL Fibrin Sealant: Non-Randomized: EVICEL is a human plasma-derived fibrin sealant composed of two components - thrombin and fibrinogen
  EVICEL Fibrin Sealant: Intraoperative (Safety Set)
Arm/Group | EVICEL Fibrin Sealant: Randomized | Standard of Care | Experimental: EVICEL Fibrin Sealant: Non-Randomized
Number analyzed (Participants) | 84 | 89 | 41
participants | 72 | 81 | 38

2. Secondary Outcome: Incidence of Adverse Events
Time Frame: up to Day 90
Measure: Number; unit: number of adverse events
Groups:
- EVICEL Fibrin Sealant: Randomized: EVICEL is a human plasma-derived fibrin sealant composed of two components - thrombin and fibrinogen.
  EVICEL Fibrin Sealant: Intraoperative (Safety Set)
- Standard of Care: Standard surgical technique for GI anastomosis. (Safety Set)
Arm/Group | EVICEL Fibrin Sealant: Randomized | Standard of Care | Experimental: EVICEL Fibrin Sealant: Non-Randomized
Number analyzed (Participants) | 84 | 89 | 41
number of adverse events | 633 | 735 | 347

3. Secondary Outcome: Incidence of GI Leak
Time Frame: 90 days
Population: The primary endpoint was absence of leak (success) within 40 days. Any data missing was considered failures. 3 EVICEL and 2 SoC subjects had missing data. These subjects were considered failures for the primary endpoint. The secondary endpoint was incidence of leak within 90 days post operatively. Missing data was not assumed to be leaks.
Measure: Number; unit: participants
Arm/Group | EVICEL Fibrin Sealant: Randomized | Standard of Care | Experimental: EVICEL Fibrin Sealant: Non-Randomized
Number analyzed (Participants) | 84 | 89 | 41
participants | 9 | 6 | 3

4. Secondary Outcome: Incidence of Stricture
Time Frame: up to Day 90
Measure: Number; unit: participants
Arm/Group | EVICEL Fibrin Sealant: Randomized | Standard of Care | Experimental: EVICEL Fibrin Sealant: Non-Randomized
Number analyzed (Participants) | 84 | 89 | 41
participants | 2 | 3 | 1

ADVERSE EVENTS:
Time Frame: AEs occurring up to study Day-90
Arm/Group | EVICEL Fibrin Sealant: Randomized | Standard of Care | Experimental: EVICEL Fibrin Sealant: Non-Randomized
Serious Adverse Events (participants affected / at risk) | 25/84 | 22/89 | 10/41
Other Adverse Events (participants affected / at risk) | 81/84 | 83/89 | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EVICEL Fibrin Sealant: Randomized (N=84) | Standard of Care (N=89) | Experimental: EVICEL Fibrin Sealant: Non-Randomized (N=41)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0 | 0
ANGINA UNSTABLE (Cardiac disorders) | 1 | 0 | 0
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 0 | 0 | 1
CARDIAC ARREST (Cardiac disorders) | 1 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0 | 0
COLITIS (Gastrointestinal disorders) | 0 | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 0 | 0
ENTEROCUTANEOUS FISTULA (Gastrointestinal disorders) | 0 | 1 | 0
ILEUS (Gastrointestinal disorders) | 3 | 2 | 0
ILEUS PARALYTIC (Gastrointestinal disorders) | 1 | 1 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1 | 0
INTESTINAL PERFORATION (Gastrointestinal disorders) | 0 | 1 | 0
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 2 | 0
SMALL INTESTINAL PERFORATION (Gastrointestinal disorders) | 0 | 1 | 1
CHEST PAIN (General disorders) | 0 | 0 | 1
PYREXIA (General disorders) | 2 | 0 | 0
PORTAL VEIN THROMBOSIS (Hepatobiliary disorders) | 0 | 1 | 0
ABDOMINAL INFECTION (Infections and infestations) | 0 | 0 | 1
ABDOMINAL SEPSIS (Infections and infestations) | 2 | 2 | 1
ABSCESS (Infections and infestations) | 0 | 1 | 0
CELLULITIS (Infections and infestations) | 0 | 1 | 0
ENDOCARDITIS (Infections and infestations) | 0 | 0 | 1
GASTROENTERITIS (Infections and infestations) | 1 | 0 | 0
HAEMATOMA INFECTION (Infections and infestations) | 1 | 0 | 0
INFECTIOUS PERITONITIS (Infections and infestations) | 2 | 0 | 0
LIVER ABSCESS (Infections and infestations) | 1 | 0 | 0
NECROTISING FASCIITIS (Infections and infestations) | 0 | 1 | 0
PELVIC ABSCESS (Infections and infestations) | 2 | 2 | 0
PERITONITIS (Infections and infestations) | 2 | 3 | 0
PYELONEPHRITIS (Infections and infestations) | 0 | 1 | 0
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 3 | 0
ANASTOMOTIC HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 1 | 0
ANASTOMOTIC LEAK (Injury, poisoning and procedural complications) | 9 | 6 | 3
ANASTOMOTIC STENOSIS (Injury, poisoning and procedural complications) | 1 | 0 | 0
INTESTINAL ANASTOMOSIS COMPLICATION (Injury, poisoning and procedural complications) | 0 | 1 | 0
POSTOPERATIVE ILEUS (Injury, poisoning and procedural complications) | 0 | 3 | 0
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0 | 0
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 0 | 1 | 0
WOUND EVISCERATION (Injury, poisoning and procedural complications) | 0 | 1 | 0
BLOOD MAGNESIUM DECREASED (Investigations) | 0 | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 1 | 0
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
URETHRAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
CRITICAL ILLNESS POLYNEUROPATHY (Nervous system disorders) | 0 | 1 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 0 | 1
DEPRESSION (Psychiatric disorders) | 1 | 0 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 | 1 | 0
URETERIC STENOSIS (Renal and urinary disorders) | 1 | 0 | 0
URETHRAL STENOSIS (Renal and urinary disorders) | 1 | 0 | 0
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1 | 0 | 0
PELVIC HAEMATOMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
BRONCHIAL SECRETION RETENTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
ABSCESS DRAINAGE (Surgical and medical procedures) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EVICEL Fibrin Sealant: Randomized (N=84) | Standard of Care (N=89) | Experimental: EVICEL Fibrin Sealant: Non-Randomized (N=41)
ANAEMIA (Blood and lymphatic system disorders) | 3 | 5 | 4
TACHYCARDIA (Cardiac disorders) | 6 | 12 | 4
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 12 | 17 | 5
ABDOMINAL PAIN (Gastrointestinal disorders) | 17 | 17 | 8
CONSTIPATION (Gastrointestinal disorders) | 14 | 17 | 11
DIARRHOEA (Gastrointestinal disorders) | 11 | 15 | 8
ILEUS (Cardiac disorders) | 6 | 5 | 1
NAUSEA (Gastrointestinal disorders) | 42 | 47 | 22
PROCTALGIA (Gastrointestinal disorders) | 3 | 5 | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 3 | 5 | 4
VOMITING (Gastrointestinal disorders) | 20 | 22 | 11
FATIGUE (General disorders) | 7 | 3 | 4
PAIN (General disorders) | 5 | 10 | 5
PYREXIA (General disorders) | 15 | 17 | 9
URINARY TRACT INFECTION (Infections and infestations) | 5 | 11 | 1
WOUND INFECTION (Infections and infestations) | 2 | 5 | 4
ANASTOMOTIC LEAK (Injury, poisoning and procedural complications) | 9 | 6 | 3
INCISION SITE PAIN (Injury, poisoning and procedural complications) | 3 | 3 | 6
PROCEDURAL PAINii (Injury, poisoning and procedural complications) | 19 | 17 | 6
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 5 | 2 | 0
C-REACTIVE PROTEIN INCREASED (Investigations) | 4 | 6 | 0
OXYGEN SATURATION DECREASED (Investigations) | 6 | 1 | 1
URINE OUTPUT DECREASED (Investigations) | 7 | 10 | 2
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 5 | 2 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 8 | 6 | 2
HYPOKALAEMIA (Metabolism and nutrition disorders) | 5 | 9 | 5
DIZZINESS (Nervous system disorders) | 5 | 9 | 4
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 3 | 5 | 2
ANXIETY (Psychiatric disorders) | 5 | 3 | 2
INSOMNIA (Psychiatric disorders) | 7 | 7 | 6
DYSURIA (Renal and urinary disorders) | 3 | 5 | 2
URINARY RETENTION (Renal and urinary disorders) | 3 | 5 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 2
PRURITUS (Skin and subcutaneous tissue disorders) | 9 | 8 | 6
HYPERTENSION (Vascular disorders) | 4 | 9 | 3
HYPOTENSION (Vascular disorders) | 13 | 16 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days